CLINICAL TRIAL: NCT06383234
Title: REduced Pain After Bariatric Surgery - Sleeve Gastrectomy
Acronym: REPABS-SG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Vincenzo Bruni, Principal Invesigator, Fondazione Policlinico Universitario Campus Bio-Medico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PAR 89/21
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Pain; Postoperative Pain; Acute Pain; Analgesia; Bariatric Surgery Candidate; Anesthesia
MeSH Terms: conditions — Pain; Pain, Postoperative; Acute Pain; Agnosia | interventions — Anesthetics, Local; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LG-TAP (Experimental): The laparoscopic guided TAP Block was performed at the beginning of surgery, injecting 15 ml of Ropivacaine Hydrochloride 0.5% on each side, using an atraumatic needle (10/15 cm length, 20 Gauge diameter) close to the anterior axillary line, between the iliac crest and the subcostal margin. Correct needle tip positioning between the transverse muscle of the abdomen and the internal oblique was verified through laparoscopic guidance.
  Interventions: Procedure: LG-TAP block with local anesthetic; Procedure: Port site infiltration
- SALINE (Placebo Comparator): The laparoscopic guided TAP Block was performed at the beginning of surgery, injecting 15 ml of Saline solution (NaCl 0.9%) on each side, using an atraumatic needle (10/15 cm length, 20 Gauge diameter) close to the anterior axillary line, between the iliac crest and the subcostal margin. Correct needle tip positioning between the transverse muscle of the abdomen and the internal oblique was verified through laparoscopic guidance.
  Interventions: Procedure: LG-TAP block with saline solution; Procedure: Port site infiltration

INTERVENTIONS:
Procedure: LG-TAP block with local anesthetic — The laparoscopic guided TAP Block was performed by surgeon at the beginning of surgery, injecting 15 ml of Ropivacaine 0.5% on each side, using an atraumatic needle (10/15 cm length, 20 Gauge diameter) close to the anterior axillary line, between the iliac crest and the subcostal margin. Correct needle tip positioning between the transverse muscle of the abdomen and the internal oblique was verified through laparoscopic guidance.
  Arms: LG-TAP
Procedure: LG-TAP block with saline solution — The laparoscopic guided TAP Block was performed by surgeon at the beginning of surgery, injecting 15 ml of Saline solution (NaCl 0.9%) on each side, using an atraumatic needle (10/15 cm length, 20 Gauge diameter) close to the anterior axillary line, between the iliac crest and the subcostal margin. Correct needle tip positioning between the transverse muscle of the abdomen and the internal oblique was verified through laparoscopic guidance.
  Arms: SALINE
Procedure: Port site infiltration — Prior the surgical incision, an infiltration of the laparoscopic access using a total of 10 ml Ropivacaine 0.5% was performed by surgeon

SUMMARY:
This study aims to analyze the effect of laparoscopic guided transversus abdominis plane (LG-TAP) block compared to placebo for postoperative analgesia following laparoscopic sleeve gastrectomy. One group of participants received a (LG-TAP) block with local anesthetic while the other group received (LG-TAP) block with saline solution (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Elective Laparoscopic Sleeve Gastrectomy
* Body Mass Index (BMI) > 35 kg/m² and at least one condition related to obesity (e.g., hypertension, type II diabetes, dyslipidemia, hepatic steatosis, etc)
* BMI > 40 kg/m², even in the absence of comorbidities
* ASA physical status score < 4

Exclusion Criteria:

* ASA physical status score ≥ 4
* Patient's refusal or inability to sign the informed consent
* Allergies to any drug provided by the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Pain Score | 24 hours
  A numerical rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain) will be used to evaluate pain at rest during 24 hours after surgery

SECONDARY OUTCOMES:
Morphine Consumption | 24 hours
  Total of intravenous morphine (expressed in milligrams) administered administered during the first 24 hours after surgery
Toradol Consumption | 24 hours
  Total of intravenous toradol (expressed in milligrams) administered administered during the first 24 hours after surgery
Nausea and/or vomiting | 48 hours
  Incidence of nausea and/or vomiting
Lenght of Hospital Stay | 72 hours
  Time between surgery and dismission from the hospital
Time to walking | 72 hours
  Time between surgery and patient starting to walk
Time to first flatus | 72 hours
  Time between surgery and patient having flatus
Surgical Complication | 7 days
  Incidence of complications related to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Bruni, MD, Principal Investigator — Fondazione Policlinico Universitario Campus Bio-Medico
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-medico, Rome, Italy

REFERENCES:
- [Background] Mongelli F, Marengo M, Bertoni MV, Volonte F, Ledingham NS, Garofalo F. Laparoscopic-Assisted Transversus Abdominis Plane (TAP) Block Versus Port-Site Infiltration with Local Anesthetics in Bariatric Surgery: a Double-Blind Randomized Controlled Trial. Obes Surg. 2023 Nov;33(11):3383-3390. doi: 10.1007/s11695-023-06825-7. Epub 2023 Sep 23. PMID 37740830
- [Result] Ripolles-Melchor J, Sanchez-Santos R, Abad-Motos A, Gimeno-Moro AM, Diez-Remesal Y, Jove-Albores P, Arago-Chofre P, Ortiz-Sebastian S, Sanchez-Martin R, Ramirez-Rodriguez JM, Trullenque-Juan R, Valenti-Azcarate V, Ramiro-Ruiz A, Correa-Chacon OC, Batalla A, Gimeno-Grauwinkel C, Sanahuja-Blasco JM, Gonzalez-Valverde FM, Galan-Menendez P, Diez-Zapirain MJ, Vilallonga R, Zorrilla-Vaca A, Pascual-Bellosta AM, Martinez-Ubieto J, Carrascosa-Miron T, Ruiz-Escobar A, Martin-Garcia-Almenta E, Suarez-de-la-Rica A, Bausili M, Palacios-Cordoba A, Olvera-Garcia MM, Meza-Vega JA, Sanchez-Pernaute A, Abad-Gurumeta A, Ferrando-Ortola C, Martin-Vaquerizo B, Torres-Alfonso JR, Aguado-Sanchez S, Sanchez-Cabezudo-Noguera F, Garcia-Erce JA, Aldecoa C; POWER 3 Study Investigators Group. Higher Adherence to ERAS Society(R) Recommendations is Associated with Shorter Hospital Stay Without an Increase in Postoperative Complications or Readmissions in Bariatric Surgery: the Association Between Use of Enhanced Recovery After Surgery Protocols and Postoperative Complications after Bariatric Surgery (POWER 3) Multicenter Observational Study. Obes Surg. 2022 Apr;32(4):1289-1299. doi: 10.1007/s11695-022-05949-6. Epub 2022 Feb 10. PMID 35143011